CLINICAL TRIAL: NCT02704702
Title: A Clinical Trial to Evaluate the Pharmacokinetics and Safety of Fimasartan and Rosuvastatin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BR-FRC-CT-102; CA16652 (Other: Celerion)
Record Dates: First submitted 2016-03-04; First posted 2016-03-10 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-02

CONDITIONS: Hypertension
Keywords: Fimasartan
MeSH Terms: conditions — Hypertension | interventions — fimasartan; Rosuvastatin Calcium

ARMS (6):
- Sequence 1 (ABC) (Other): Period 1(Treatment A) → Period 2(Treatment B) → Period 3(Treatment C)
  There will be a washout of at least 7 days between the each period.
  Interventions: Drug: Fimasartan; Drug: Rosuvastatin; Drug: Fimasartan + Rosuvastatin
- Sequence 2 (ACB) (Other): Period 1(Treatment A) → Period 2(Treatment C) → Period 3(Treatment B)
  There will be a washout of at least 7 days between the each period.
  Interventions: Drug: Fimasartan; Drug: Rosuvastatin; Drug: Fimasartan + Rosuvastatin
- Sequence 3 (BAC) (Other): Period 1(Treatment A) → Period 2(Treatment B) → Period 3(Treatment 3)
  There will be a washout of at least 7 days between the each period.
  Interventions: Drug: Fimasartan; Drug: Rosuvastatin; Drug: Fimasartan + Rosuvastatin
- Sequence 4 (BCA) (Other): Period 1(Treatment B) → Period 2(Treatment C) → Period 3(Treatment A)
  There will be a washout of at least 7 days between the each period.
  Interventions: Drug: Fimasartan; Drug: Rosuvastatin; Drug: Fimasartan + Rosuvastatin
- Sequence 5 (CAB) (Other): Period 1(Treatment C) → Period 2(Treatment A) → Period 3(Treatment B)
  There will be a washout of at least 7 days between the each period.
  Interventions: Drug: Fimasartan; Drug: Rosuvastatin; Drug: Fimasartan + Rosuvastatin
- Sequence 6 (CBA) (Other): Period 1(Treatment C) → Period 2(Treatment B) → Period 3(Treatment A)
  There will be a washout of at least 7 days between the each period.
  Interventions: Drug: Fimasartan; Drug: Rosuvastatin; Drug: Fimasartan + Rosuvastatin

INTERVENTIONS:
Drug: Fimasartan
Drug: Rosuvastatin
Drug: Fimasartan + Rosuvastatin

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of Fimasartan and rosuvastatin when coadministered or administered alone as a single dose or as multiple doses to healthy male subjects.

DETAILED DESCRIPTION:
This is an open-label, randomized, 6-sequence, 3-period, 3-way crossover study. Within each period, randomized subjects will be 2 dosing regimens with the same drug(fimasartan or rosuvastatin) or study drug combination(fimasartan+rosuvastatin) on day 1 and quaque die(qd) from day 4 to day 10. After day 1 and day 10 dosing will be followed by pharmacokinetic sampling for 48 hours or 72 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian male 19-55 years of age.
2. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2 at screening.
3. Medically healthy with no clinically significant medical history.
4. Understands the study procedures in the Informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. History or presence of clinically significant medical or psychiatric condition or disease.
2. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
3. Seated blood pressure is less than 90/60 mmHg or greater than 140/90 mmHg at screening.
4. Plasma donation within 7 days prior to the first dose of study drug.
5. Participation in another clinical trial within 28 days prior to the first dose of study drug(s).

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Sterling, M.D, Principal Investigator — Celelion, Inc.

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1 (ABC): Period 1(Treatment A) → Period 2(Treatment B) → Period 3(Treatment C)
  There will be a washout of at least 7 days between the each period.
  Fimasartan
  Rosuvastatin
  Fimasartan + Rosuvastatin
- Sequence 2 (ACB): Period 1(Treatment A) → Period 2(Treatment C) → Period 3(Treatment B)
  There will be a washout of at least 7 days between the each period.
  Fimasartan
  Rosuvastatin
  Fimasartan + Rosuvastatin
- Sequence 3 (BAC): Period 1(Treatment A) → Period 2(Treatment B) → Period 3(Treatment 3)
  There will be a washout of at least 7 days between the each period.
  Fimasartan
  Rosuvastatin
  Fimasartan + Rosuvastatin
- Sequence 4 (BCA): Period 1(Treatment B) → Period 2(Treatment C) → Period 3(Treatment A)
  There will be a washout of at least 7 days between the each period.
  Fimasartan
  Rosuvastatin
  Fimasartan + Rosuvastatin
- Sequence 5 (CAB): Period 1(Treatment C) → Period 2(Treatment A) → Period 3(Treatment B)
  There will be a washout of at least 7 days between the each period.
  Fimasartan
  Rosuvastatin
  Fimasartan + Rosuvastatin
- Sequence 6 (CBA): Period 1(Treatment C) → Period 2(Treatment B) → Period 3(Treatment A)
  There will be a washout of at least 7 days between the each period.
  Fimasartan
  Rosuvastatin
  Fimasartan + Rosuvastatin
Period: Overall Study
Arm/Group | Sequence 1 (ABC) | Sequence 2 (ACB) | Sequence 3 (BAC) | Sequence 4 (BCA) | Sequence 5 (CAB) | Sequence 6 (CBA)
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 5 | 6 | 6 | 5 | 4 | 4
Not Completed | 1 | 0 | 0 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 2 (ACB) | Sequence 3 (BAC) | Sequence 1 (ABC) | Sequence 4 (BCA) | Sequence 5 (CAB) | Sequence 6 (CBA) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 36
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 5 | 6 | 5 | 6 | 6 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 6 | 6 | 36
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve
Description: This Outcome is the Area Calculated using the Linear Trapezoidal with Linear Interpolation Method
Time Frame: For Fimasartan PK(Treatment A and C) : Post-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24, 36, 48 in each period/For Rosuvastatin PK(Treatment B and C) : Post-dose, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 48, 72 in each period
Measure: Geometric Mean (95% Confidence Interval); unit: ng*hr/mL
Groups:
- Treatment A(Single Dose); Treatment A(Multiple Dose); Treatment B(Single Dose); Treatment B(Multiple Dose); Treatment C(Single Dose_Fimasartan); Treatment C(Single Dose_Rosuvastatin); Treatment C(Multiple Dose_Fimasartan); Treatment C(Multiple Dose_Rosuvastatin): Sequence 1(ABC)/Sequence 2(ACB)/Sequence 3(BAC)/Sequence 4(BCA)/Sequence 5(CAB)/Sequence 6(CBA)
  There will be a washout of at least 7 days between the each period.
  Treatment A: Fimasartan
  Treatment B: Rosuvastatin
  Treatment C: Fimasartan + Rosuvastatin
Arm/Group | Treatment A(Single Dose) | Treatment A(Multiple Dose) | Treatment B(Single Dose) | Treatment B(Multiple Dose) | Treatment C(Single Dose_Fimasartan) | Treatment C(Single Dose_Rosuvastatin) | Treatment C(Multiple Dose_Fimasartan) | Treatment C(Multiple Dose_Rosuvastatin)
Number analyzed (Participants) | 34 | 32 | 35 | 32 | 34 | 34 | 34 | 34
ng*hr/mL | 690.43 [645.39 to 809.51] | 820.86 [757.50 to 980.63] | 86.442 [82.210 to 105.59] | 114.55 [106.95 to 138.50] | 702.20 [653.05 to 830.43] | 85.078 [78.638 to 115.45] | 880.19 [819.63 to 1018.7] | 98.957 [91.971 to 120.50]

2. Primary Outcome: Maximum Observed Concentration
Description: This Outcome is the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated.
Time Frame: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Treatment A(Single Dose) | Treatment A(Multiple Dose) | Treatment B(Single Dose) | Treatment B(Multiple Dose) | Treatment C(Single Dose_Fimasartan) | Treatment C(Multiple Dose_Fimasartan) | Treatment C(Single Dose_Rosuvastatin) | Treatment C(Multiple Dose_Rosuvastatin)
Number analyzed (Participants) | 34 | 32 | 35 | 32 | 34 | 34 | 34 | 34
ng/mL | 289.12 [272.28 to 373.86] | 362.14 [339.10 to 523.63] | 9.305 [8.755 to 11.733] | 11.706 [10.927 to 14.416] | 283.73 [268.35 to 383.63] | 341.92 [329.13 to 462.35] | 12.581 [11.697 to 17.502] | 13.687 [12.713 to 17.300]

3. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration
Description: This Outcome is the time it takes a drug to reach Cmax
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | Treatment A(Single Dose) | Treatment A(Multiple Dose) | Treatment B(Single Dose) | Treatment B(Multiple Dose) | Treatment C(Single Dose_Fimasartan) | Treatment C(Multiple Dose_Fimasartan) | Treatment C(Single Dose_Rosuvastatin) | Treatment C(Multiple Dose_Rosuvastatin)
Number analyzed (Participants) | 34 | 32 | 36 | 32 | 34 | 34 | 34 | 34
hr | 0.749 [0.50 to 2.00] | 0.635 [0.49 to 2.51] | 2.999 [1.00 to 5.03] | 4.505 [1.01 to 5.06] | 0.750 [0.50 to 1.50] | 0.751 [0.50 to 4.00] | 2.003 [1.00 to 5.00] | 1.506 [1.00 to 5.09]

ADVERSE EVENTS:
Time Frame: Participants assessed 13 days for each intervention, a total of approximately 4 weeks
Description: Safety population included all population who receive at least 1 dose of study drug
Groups:
- Treatment B(Multiiple Dose); Treatment C(Single Dose); Treatment C(Multiple Dose): Sequence 1(ABC)/Sequence 2(ACB)/Sequence 3(BAC)/Sequence 4(BCA)/Sequence 5(CAB)/Sequence 6(CBA)
  There will be a washout of at least 7 days between the each period.
  Treatment A: Fimasartan
  Treatment B: Rosuvastatin
  Treatment C: Fimasartan + Rosuvastatin
Arm/Group | Treatment A(Single Dose) | Treatment A(Multiple Dose) | Treatment B(Single Dose) | Treatment B(Multiiple Dose) | Treatment C(Single Dose) | Treatment C(Multiple Dose)
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/33 | 0/35 | 0/34 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/35 | 1/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 2/34 | 6/33 | 6/35 | 7/34 | 6/34 | 8/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A(Single Dose) (N=34) | Treatment A(Multiple Dose) (N=33) | Treatment B(Single Dose) (N=35) | Treatment B(Multiiple Dose) (N=34) | Treatment C(Single Dose) (N=34) | Treatment C(Multiple Dose) (N=34)
Thoracic vertebral fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — It is resulted in discontinuation from the study. Approximately 3.4 days following dosing with rosuvastatin 20mg alone, the subject was cutting a tree branch when the branch fell on top of him and he was transported to the hospital via ambulance.
Right clavicle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right radius fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
multiple closed rib fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Right sided pneumothorax (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A(Single Dose) (N=34) | Treatment A(Multiple Dose) (N=33) | Treatment B(Single Dose) (N=35) | Treatment B(Multiiple Dose) (N=34) | Treatment C(Single Dose) (N=34) | Treatment C(Multiple Dose) (N=34)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Several sampling time deviations occurred during the clinical conduct of this study. Actual sampling times relative to dosing time were used for caculation of PK parameters.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Obligation of disclosure restriction continue for 3 years from the date of termination or expiration of Agreement effected on November 16th, 2015.